CLINICAL TRIAL: NCT05939973
Title: A Feasibility Study Examining Safety and Preliminary Effectiveness of a Procedural Technique Using an Endoscopic Suturing Device (g-Cath EZ Delivery Catheter With Snowshoe Suture Anchors) and Associated Devices for the Treatment of Primary Obesity
Brief Title: A Feasibility Study for the Treatment of Primary Obesity Cross-over Arm
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: USGI Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 50598 TPR
Record Dates: First submitted 2023-06-23; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-06

CONDITIONS: Obesity, Primary
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: This is a multi-center, open-label, cross-over arm from the 2-group randomized pilot study evaluating a treatment for obesity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Crossover (Other): Continuation of POSE2.0 expansion study evaluating the safety and preliminary effectiveness of the Pose 2 procedure using the g-Cath EZ Suture Anchor Delivery Catheter as a primary weight loss intervention in the control arm, defined as crossover subjects from POSE2.0 Expansion Study.
  Interventions: Device: g-Cath EZ Delivery Catheter with Snowshoe Suture Anchors

INTERVENTIONS:
Device: g-Cath EZ Delivery Catheter with Snowshoe Suture Anchors — The intent is to evaluate the safety and preliminary efficacy of a new Snowshoe suture placement pattern, POSE2.0 (sutures placed in the mid + distal body without fundus), with a moderate intensity diet and exercise program.

SUMMARY:
Cross-over arm of the pilot study evaluating a treatment for obesity.

DETAILED DESCRIPTION:
This is a multi-center, open-label, cross-over arm from the 2-group randomized pilot study evaluating a treatment for obesity. The intent is to evaluate the safety and preliminary efficacy of a new Snowshoe suture placement pattern, POSE2.0 (sutures placed in the mid + distal body without fundus), with a moderate intensity diet and exercise program. The procedure will be performed using the g-Cath EZ Delivery Catheter with Snowshoe Suture Anchors (AKA g-Cath or g-Cath EZ) and associated devices (g-Prox EZ, g-Lix and Transport), known collectively as the Incisionless Operating Platform (IOP). Efficacy will be evaluated based on changes in weight loss through 12 months. Adverse events will be recorded throughout the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Subject agrees to be compliant with study requirements and adhere to post-operative dietary & exercise recommendations for the duration of the study.
3. Subjects between the ages of 22-60 years.
4. If female, be either post-menopausal, surgically sterile, or agree to practice birth control during year of study and have negative serum HCG at screening/baseline.
5. Met BMI inclusion criteria when enrolled in the study as defined by a Body Mass Index (BMI) of ≥ 35 and < 40 with one or more obesity related co-morbid conditions (defined by 1991 NIH Guidelines (Appropriateness Criteria for Bariatric Surgery: Beyond the NIH Guidelines).

   1. Pre-diabetes - Fasting plasma glucose test >100 mg/dl but ≤125 or oral glucose tolerance test ≥140 mg/dl but <200.
   2. Diabetes - Individuals taking insulin and/or oral hypoglycemic medications or have a fasting glucose >126 mg/dl.
   3. Hypertension - SBP>140 or DBP>90 or the use of an antihypertensive medication.
   4. Dyslipidemia - Triglycerides > 250 mg/dl or cholesterol > 220 mg/dl or HDL < 35 mg/dl or LDL > 200 or use of lipid lowering medications.
   5. Sleep Apnea - A formal sleep study test consistent with this diagnosis; Epworth sleepiness scale ≥ 6; Polysomnography with respiratory disturbance index ≥ 10 hyponeic and/or apneic episodes per hour of sleep.
   6. Venous Stasis Disease - Presence or history of pretibial venous stasis ulcers.
   7. Chronic Joint Disease - Deterioration of joint cartilage and the formation of new bone (bone spurs) at the margins of the joints.
6. Absence of current severe systemic disease (including, but not limited to: coronary artery disease, chronic obstructive pulmonary disease, congestive heart failure, cancer, and chronic renal disease).
7. Agrees not to undergo any additional weight loss interventional procedures or liposuction for 12 months following study enrollment.
8. Have not taken any prescription or over the counter weight loss medications OR those that can suppress appetite/induce weight loss for at least 6 months and agrees not to utilize for 12 months following study enrollment (including all stimulant medication).
9. Subjects must be willing to possibly forego any future weight loss procedures (i.e. Vertical Sleeve Gastrectomy) given the unknown long-term effects.
10. Residing within a reasonable distance from the Investigator's treating office (~50 miles) and willing and able to travel to the Investigator's office to complete all routine follow-up visits.

Exclusion Criteria:

1. History of (or intra-operative evidence of) prior bariatric, gastric or esophageal surgery.
2. Esophageal stricture or other anatomy and/or condition that could preclude passage of endoluminal instruments or procedure execution.
3. Moderate gastro-esophageal reflux disease (GERD), defined as symptoms that cause subject severe discomfort, compromise performance of daily activities, and/or condition is not entirely controlled with drug therapy.
4. Large hiatal hernia (>3 cm) by history or as determined by pre-enrollment endoscopy.
5. Pancreatic insufficiency/disease.
6. History of gastroparesis or symptoms that would be suggestive of gastroparesis or generalized dysmotility (e.g. esophago-gastric motility issues and lower esophageal sphincter abnormalities).
7. Pregnancy or plans of pregnancy in the next 12 months.
8. History of a known diagnosis or pre-existing symptom of rheumatoid arthritis, scleroderma, system lupus, or other autoimmune connective tissue disorder.
9. Immunosuppressive medications or systemic steroids (i.e., oral prednisone) within 6 months of Visit 1. Intranasal/inhaled steroids are acceptable.
10. Unable or unwilling to avoid use of aspirin and/or non-steroidal anti-inflammatory drugs (NSAIDs), or other medications known to be gastric irritants beginning two weeks prior to enrollment and throughout the entire study.
11. History of inflammatory disease of the GI tract; coagulation disorders; hepatic insufficiency or cirrhosis.
12. Active gastric erosion, lesion, or gastric/duodenal ulcer.
13. History of or current platelet or coagulation dysfunction, such as hemophilia.
14. History or present use of insulin or insulin derivatives for treatment of diabetes.
15. Type II Diabetes Mellitus (as defined by HgbA1c >6.5%) for greater than 11 years at the time of enrollment.
16. If smoker, plans to quit smoking in the year after enrollment.
17. Portal hypertension and/or varices.
18. Patient has a history of drug or alcohol abuse or positive at screening for drugs of abuse.
19. Patient is currently using marijuana/cannabis for either medicinal or recreational use, or has plans to start using over the next 12 months.
20. Present or history of psychosis, bipolar disease, or obsessive-compulsive disorder after pre-enrollment history and medical /psychological assessment.
21. Beck Depression Inventory (Short) Score ≥ 12 and/or uncontrolled depression after pre-enrollment psychological and medical assessment. 1
22. Patient score >2 in any of the 9 identified symptoms on the Gastroparesis Cardinal Symptom Index (GCSI)
23. Patient with a 13C-Spirulina Gastric Emptying Breath Test (GEBT) result that is less than a kPCD/min of 34.4 at 120 minutes or 43 at 180 minutes
24. Non-ambulatory or has significant impairment of mobility (i.e. cannot ambulate for 30 minutes).
25. Known hormonal or genetic cause for obesity including untreated hypothyroidism (TSH >5.0 U/ml).
26. Participating in another clinical study that would conflict with the requirements of the study protocol as described.
27. Subjects with a personal history of allergic/anaphylactic reactions including hypersensitivity to the drugs or materials that will be utilized in the study procedure.
28. Physician's assessment that the subject is not an appropriate candidate.

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Mean Percent TBWL at 3 months | 3 months.
  Mean Percent TBWL at 3 months.
Mean Percent TBWL at 12 months | 12 months.
  Mean Percent TBWL at 12 months.
Percentage of subjects with ≥5% TBWL at 3 months | 3 months.
  Percentage of subjects with ≥5% TBWL at 3 months.
Percentage of subjects with ≥5% TBWL at 12 months | 12 months.
  Percentage of subjects with ≥5% TBWL at 12 months.
Overall incidence of device and procedure related adverse events through 12 months | 12 months
  Overall incidence of device and procedure related adverse events through 12 months.

SECONDARY OUTCOMES:
To investigate observational efficacy objectives of the POSE2.0 procedure | Change from baseline at 3 months
  Change from baseline at 3 months in Percent EWL
To investigate observational efficacy objectives of the POSE2.0 procedure | Change from baseline at 12 months
  Change from baseline at 12 months in Percent EWL
To investigate observational efficacy objectives of the POSE2.0 procedure | Change from baseline at 3 months
  Change from baseline at 3 months in BMI reduction
To investigate observational efficacy objectives of the POSE2.0 procedure | Change from baseline at 12 months
  Change from baseline at 12 months in BMI reduction
To investigate observational efficacy objectives of the POSE2.0 procedure | Change from baseline at 3 months
  Change from baseline at 3 months in weight loss (lb/kg)
To investigate observational efficacy objectives of the POSE2.0 procedure | Change from baseline at 12 months
  Change from baseline at 12 months in weight loss (lb/kg)
To investigate observational efficacy objectives of the POSE2.0 procedure | Change from baseline at 3 months
  Change from baseline at 3 months in waist circumference
To investigate observational efficacy objectives of the POSE2.0 procedure | Change from baseline at 12 months
  Change from baseline at 12 months in waist circumference
Change from baseline at 12 months in Quality of Life Scores | Change from baseline at 12 months
  The IWQOL-Lite questionnaire is a validated, 31-item, self-report measure of obesity-specific quality of life. In addition to a total score, there are scores on five domains: Physical function; Self-esteem; Sexual life; Public distress; Work.
Change from baseline at 12 months in Co-morbidities | Change from baseline at 12 months
  Change from baseline at 12 months in Co-morbidities.
Change from baseline at 12 months in liver function | Change from baseline at 12 months
  Liver function panel will be administered at baseline and at 12 months to assess change in liver function.

CONTACTS AND LOCATIONS:
Overall Officials: Barham Abu Dayyeh, MD, MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No